CLINICAL TRIAL: NCT05669898
Title: Multimodal Analgesia for Unilateral Total Knee Arthroplasty: Impact of Continuous Adductor Canal Infusion Combined With NSAID vs. Intravenous Morphine Patient-controlled Analgesia Combined With Single-injection Adductor Canal Block
Brief Title: Continuous Adductor Canal Infusion vs. Single-injection Adductor Canal Block for Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPEVGH IRB No.: 2018-08-007A
Record Dates: First submitted 2022-05-23; First posted 2023-01-03 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Arthroplasty, Replacement, Knee; Pain, Postoperative; Multimodal Analgesia
Keywords: Arthroplasty, Replacement, Knee; Regional analgesia; multimodal analgesia; Rehabilitation; Recovery of Function
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A two-arm parallel assignment involves two groups of participants receiving multimodal analgesia after unilateral total knee arthroplasty. One group receives a single-injection adductor canal block combined with intravenous morphine patient-controlled analgesia, and the other group receives continuous adductor canal infusion in combination with intermittent intravenous non-steroidal anti-inflammatory drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-injection ACB combined with IV-PCA morphine (Active Comparator): Allocation of which participant is to receive single-injection adductor canal block combined with intravenous morphine patient-controlled analgesia (IV-morphine PCA) is determined by randomization, using a computer-generated random sequence and opaque sealed envelopes. After completion of the TKA surgery and surgical suturing, adductor canal block will be performed by an anesthesiologist. Under ultrasound guidance, the femoral artery and the saphenous nerve are identified in the middle one-third of the thigh, deep to the sartorious muscle in the adductor canal. The sartorious and adductor muscles form the roof and the floor of the canal, respectively. Following skin infiltration, 20 mL of 0.25% bupivacaine with 1:400000 epinephrine is injected through a 3-inch, 23-gauge, short bevel block needle. Finally, the IV-morphine PCA will be connected to the intravenous catheter of the patient for postoperative pain management.
  Interventions: Behavioral: Pain scores (numerical rating scale at rest and motion): will be assessed with numerical rating scale at both rest and motion on both knees.; Other: Brief Pain Inventory (Short Form), WOMAC Osteoarthritis index, and Lower extremity functional scale; Behavioral: Rehabilitation physiotherapy
- Continuous adductor canal infusion combined with intravenous NSAID (Active Comparator): Allocation of which participant is to receive continuous adductor canal infusion in combination with intermittent intravenous non-steroidal anti-inflammatory drug (NSAID) is determined by randomization, using a computer-generated random sequence and opaque sealed envelopes. After completion of the TKA surgery and surgical suturing, a peripheral nerve catheter will be implanted into adductor canal by an anesthesiologist. Under ultrasound guidance, the femoral artery and the saphenous nerve are identified in the middle one-third of the thigh, deep to the sartorious muscle in the adductor canal. The sartorious and adductor muscles form the roof and the floor of the canal, respectively. Following the peripheral nerve catheter is implanted, 20 mL of 0.25% bupivacaine with 1:400000 epinephrine is injected through the catheter. Intravenous tenoxicam 20 mg for a total amount of 3 doses at 24-hour interval after surgery will be added in the postoperative pain management.
  Interventions: Behavioral: Pain scores (numerical rating scale at rest and motion): will be assessed with numerical rating scale at both rest and motion on both knees.; Other: Brief Pain Inventory (Short Form), WOMAC Osteoarthritis index, and Lower extremity functional scale; Behavioral: Rehabilitation physiotherapy

INTERVENTIONS:
Behavioral: Pain scores (numerical rating scale at rest and motion): will be assessed with numerical rating scale at both rest and motion on both knees. — Pain scores will be assessed with numerical rating scale at both rest and motion on both knees.
Other: Brief Pain Inventory (Short Form), WOMAC Osteoarthritis index, and Lower extremity functional scale — For the functional assessment both before and after TKA surgery.
Behavioral: Rehabilitation physiotherapy — Rehabilitation physiotherapy will be assessed with knee range of motion (both active and maximal passive), muscle power at abduction and adduction, single leg stance test, six-minute walk test for assessment of the functional recovery of both knees.

SUMMARY:
Multimodal analgesia (MMA) has been endorsed to improve postoperative analgesia and functional activity after surgery, and integrating regional analgesia to reduce the consumption of opioid has also been used in postoperative pain management. The investigator try to find a better combination of MMA for postoperative analgesia and functional recovery for patients receiving TKA in Taiwan, therefore the effect of single-injection and continuous infusion of peripheral nerve block is compared in patient undergoing unilateral TKA. The investigators hypothesize that continuous adductor canal infusion is as effective as single-injection adductor canal block for postoperative pain relief under intravenous PCA after TKA surgery. Based on that, the investigators conduct this prospective, randomized controlled trial to examine our hypothesis.

DETAILED DESCRIPTION:
The study compares the effect of two multimodal analgesia protocols, the one integrating IVPCA morphine with single-injection adductor canal block and the other integrating continuous adductor canal infusion with timely administered intravenous tenoxicam, on postoperative analgesia and functional activity after TKA. To assess the outcome of both modalities, The investigators can have more comparative result of pain score and other functional parameters like range of motion of knee joint and muscle strength. Based on that, the investigators try to find a better multimodal analgesic approach for postoperative analgesia and functional recovery for patients receiving TKA in Taiwan. The investigators hypothesize that multimodal analgesia using continuous adductor canal infusion and intravenous tenoxicam are as effective as another modality using IVPCA and single-injection adductor canal block for postoperative pain relief after TKA surgery. However, continuous adductor canal infusion integrated with intravenous tenoxicam might reduce the occurrence of opioid-related side effect and enhance the functional recovery. Based on that, the investigators conduct this prospective, randomized controlled trial to examine our hypothesis.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of knee osteoarthritis
* Must be aged between 20 to 90 years old
* Must be scheduled for unilateral total knee arthroplasty surgery
* Must agree to enroll into the clinical trial and have signed the written informed consent

Exclusion Criteria:

* American Society of Anesthesiologists physical status class IV-V
* Elevated liver enzymes or liver failure
* Renal dysfunction (serum creatinine level ≥ 1.5 mg/dL)
* Cardiac failure
* Organ transplantation recipient
* Stroke
* Major neurological deficit with lower extremity muscle weakness
* Sensory and motor disorders in lower limb
* Coagulopathy or thrombocytopenia
* Previous drug dependency
* Patients who used illicit drugs within six months
* Chronic use of opioids
* Allergy to local anesthetics and drug used in experiment
* Inability to walk independently
* Inability to comprehend pain assessment
* Refusal for implanting a continuous peripheral nerve catheter
* Refusal for enrolling in study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain scores at rest and motion | Baseline (day of admission)
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.
Change in Pain scores at rest and motion | Hour 2 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.
Change in Pain scores at rest and motion | Hour 8 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.
Change in Pain scores at rest and motion | Hour 24 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.
Change in Pain scores at rest and motion | Hour 36 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.
Change in Pain scores at rest and motion | Hour 48 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.
Change in Pain scores at rest and motion | Hour 60 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.
Change in Pain scores at rest and motion | Hour 72 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.
Change in Pain scores at rest and motion | 1 day of discharge
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.
Change in Pain scores at rest and motion | Month 3 after surgery
  Assess the pain intensity with numerical rating scale both at rest and motion in each knee. A 11 point (0-10) numerical rating scale defines 0 as no pain and 10 as the worst pain imaginable.

SECONDARY OUTCOMES:
Rehabilitation physiotherapy: Knee flexion angle | Baseline (day of admission)
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Rehabilitation physiotherapy: Knee flexion angle | Hour 24 after surgery
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Rehabilitation physiotherapy: Knee flexion angle | Hour 72 after surgery
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Rehabilitation physiotherapy: Knee flexion angle | 1 Day of discharge
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Rehabilitation physiotherapy: Knee flexion angle | Month 3 after surgery
  Maximal range of motion at both continuous passive motion and active motion will be assessed with protractor (degrees)
Rehabilitation physiotherapy: knee muscle strength | Baseline (day of admission)
  Muscle power of the surgical knee at abduction and adduction accessed by JTech Commander Echo Manual Muscle Tester
Rehabilitation physiotherapy: knee muscle strength | Hour 24 after surgery
  Muscle power of the surgical knee at abduction and adduction accessed by JTech Commander Echo Manual Muscle Tester
Rehabilitation physiotherapy: knee muscle strength | Hour 72 after surgery
  Muscle power of the surgical knee at abduction and adduction accessed by JTech Commander Echo Manual Muscle Tester
Rehabilitation physiotherapy: knee muscle strength | 1 day of discharge
  Muscle power of the surgical knee at abduction and adduction accessed by JTech Commander Echo Manual Muscle Tester
Rehabilitation physiotherapy: knee muscle strength | Month 3 after surgery
  Muscle power of the surgical knee at abduction and adduction accessed by JTech Commander Echo Manual Muscle Tester
Rehabilitation physiotherapy: Six minute walk test | Baseline (day of admission)
  To assess the walk ability (6-minute walk distance) before and after surgery (meters)
Rehabilitation physiotherapy: Six minute walk test | Hour 24 after surgery
  To assess the walk ability (6-minute walk distance) before and after surgery (meters)
Rehabilitation physiotherapy: Six minute walk test | Hour 72 after surgery
  To assess the walk ability (6-minute walk distance) before and after surgery (meters)
Rehabilitation physiotherapy: Six minute walk test | 1 date of discharge
  To assess the walk ability (6-minute walk distance) before and after surgery (meters)
Rehabilitation physiotherapy: Six minute walk test | Month 3 after surgery
  To assess the walk ability (6-minute walk distance) before and after surgery (meters)
Rehabilitation physiotherapy: Single leg stance test | Baseline (day of admission)
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Rehabilitation physiotherapy: Single leg stance test | Hour 24 after surgery
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Rehabilitation physiotherapy: Single leg stance test | Hour 72 after surgery
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Rehabilitation physiotherapy: Single leg stance test | 1 day of discharge
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Rehabilitation physiotherapy: Single leg stance test | Month 3 after surgery
  To assess the stance ability and static postural and balance control on one leg without help either with eyes opened or closed before and after TKA surgery (assessed as seconds)
Functional questionnaire: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Osteoarthritis Index | Baseline (day of admission)
  For functional pain assessment
Functional questionnaire: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Osteoarthritis Index | 1 day of discharge
  For functional pain assessment
Functional questionnaire: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Osteoarthritis Index | Month 3 after surgery
  For functional pain assessment
Functional questionnaire: Brief pain inventory (BPI) short form | Baseline (day of admission)
  For functional pain assessment
Functional questionnaire: Brief pain inventory (BPI) short form | 1 day of discharge
  For functional pain assessment
Functional questionnaire: Brief pain inventory (BPI) short form | Month 3 after surgery
  For functional pain assessment
Functional questionnaire: Lower extremity functional scale | Baseline (day of admission)
  Scoring scales from 0 to 80 with the maximum score being 80 and the lower score meaning the the greater disability.
Functional questionnaire: Lower extremity functional scale | 1 date of discharge
  Scoring scales from 0 to 80 with the maximum score being 80 and the lower score meaning the the greater disability.
Functional questionnaire: Lower extremity functional scale | Month 3 after surgery
  Scoring scales from 0 to 80 with the maximum score being 80 and the lower score meaning the the greater disability.
Adverse events | Baseline (day of admission)
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 2 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 8 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 24 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 36 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 48 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 60 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Hour 72 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | 1 day of discharge
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia
Adverse events | Month 3 after surgery
  Adverse events will be assessed with items including nausea, vomiting, somnolence, dizziness, urinary retention, skin itch, respiratory depression, and lower limb weakness, numbness, and allodynia

CONTACTS AND LOCATIONS:
Overall Officials: Hsu Ma, MD, PhD, Study Chair — Institutional Review Board, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No